CLINICAL TRIAL: NCT04482166
Title: Learning Curve of Fiberoptic-guided Tracheal Intubation Through Supraglottic Airway Device for Pediatric Difficult Airway Manikin
Brief Title: Learning Curve of Fiberoptic Intubation Through Supraglottic Airway Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Clinical associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2006-160-1135
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Intubation;Difficult
Keywords: Fiberoptic bronchoscope; Supraglottic airway

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Candidates (Experimental): Training of fiberoptic-guided tracheal intubation through supraglottic airway device to pediatric airway manikin
  Interventions: Other: Training; Device: supraglottic airway device

INTERVENTIONS:
Other: Training — 20-times training of fiberoptic-guided tracheal intubation through supraglottic airway device to pediatric airway manikin
Device: supraglottic airway device — supraglottic airway device

SUMMARY:
This study aims to obtain learning curve data of residents for fiberoptic-guided tracheal intubation through supraglottic airway device for pediatric difficult airway manikin.

DETAILED DESCRIPTION:
Residents under anesthesiology training will undergo a simulation practice to a pediatric airway manikin, after a single demonstration by an expert for fiberoptic-guided tracheal intubation through supraglottic airway device. The participants will do the same practice 20 times to the same manikin.

ELIGIBILITY:
Inclusion Criteria:

* Residents under anesthesiology training with experience of more than 30 times of supraglottic airway device insertion and manipulation of fiberoptic bronchoscope

Exclusion Criteria:

* Prior experience of fiberoptic-guided tracheal intubation through supraglottic airway device
* Prior experience of training for fiberoptic-guided tracheal intubation through supraglottic airway device

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Elapsed time to succeed endotracheal intubation for each training period | From start of each training period to success of endotracheal intubation, not to exceed 10 minutes

SECONDARY OUTCOMES:
Elapsed time to successful insertion of supraglottic airway device and ventilation of the manikin for each training period | From start of each training period to success of ventilation, not to exceed 10 minutes
Elapsed time to identification of vocal cords via fiberoptic bronchoscope for each training period | From start of each training period to identification of vocal cords, not to exceed 10 minutes
Elapsed time to introduction of fiberoptic bronchoscope into the trachea for each training period | From start of each training period to introduction of fiberoptic bronchoscope into the trachea, not to exceed 10 minutes
Success rate of endotracheal intubation for each training period | From start of each training period to success of endotracheal intubation, not to exceed 10 minutes
Number of trials | From start of each training period to success of endotracheal intubation, not to exceed 10 minutes
  Number of trials to succeed ventilation, vocal cord identification, fiberoptic bronchoscope introduction, endotracheal intubation for each training period

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Hyun Lee, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Other, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stein ML, Park RS, Kovatsis PG. Emerging trends, techniques, and equipment for airway management in pediatric patients. Paediatr Anaesth. 2020 Mar;30(3):269-279. doi: 10.1111/pan.13814. Epub 2020 Feb 5. PMID 32022437
- [Background] Hunyady A, Polaner D. Pediatric airway management education and training. Paediatr Anaesth. 2020 Mar;30(3):362-370. doi: 10.1111/pan.13808. Epub 2020 Jan 16. PMID 31887239
- [Background] Black AE, Flynn PE, Smith HL, Thomas ML, Wilkinson KA; Association of Pediatric Anaesthetists of Great Britain and Ireland. Development of a guideline for the management of the unanticipated difficult airway in pediatric practice. Paediatr Anaesth. 2015 Apr;25(4):346-62. doi: 10.1111/pan.12615. Epub 2015 Feb 16. PMID 25684039
- [Background] Kovatsis PG. Continuous ventilation during flexible fiberscopic-assisted intubation via supraglottic airways. Paediatr Anaesth. 2016 Apr;26(4):457-8. doi: 10.1111/pan.12863. No abstract available. PMID 26956516
- [Background] Dalal PG, Dalal GB, Pott L, Bezinover D, Prozesky J, Bosseau Murray W. Learning curves of novice anesthesiology residents performing simulated fibreoptic upper airway endoscopy. Can J Anaesth. 2011 Sep;58(9):802-9. doi: 10.1007/s12630-011-9542-2. Epub 2011 Jun 28. PMID 21710368
- [Background] Altun D, Ozkan-Seyhan T, Camci E, Sivrikoz N, Orhan-Sungur M. Learning Curves for Two Fiberscopes in Simulated Difficult Airway Scenario With Cumulative Sum Method. Simul Healthc. 2019 Jun;14(3):163-168. doi: 10.1097/SIH.0000000000000368. PMID 30908421
- [Background] Oliveira KF, Arzola C, Ye XY, Clivatti J, Siddiqui N, You-Ten KE. Determining the amount of training needed for competency of anesthesia trainees in ultrasonographic identification of the cricothyroid membrane. BMC Anesthesiol. 2017 Jun 2;17(1):74. doi: 10.1186/s12871-017-0366-7. PMID 28577552
- [Background] Orhan-Sungur M, Altun D, Ozkan-Seyhan T, Aygun E, Koltka K, Camci E. Learning curve of ultrasound measurement of subglottic diameter for endotracheal tube selection in pediatric patients. Paediatr Anaesth. 2019 Dec;29(12):1194-1200. doi: 10.1111/pan.13751. Epub 2019 Oct 20. PMID 31583796
- [Background] Kim HJ, Park HS, Kim SY, Ro YJ, Yang HS, Koh WU. A Randomized Controlled Trial Comparing Ambu AuraGain and i-gel in Young Pediatric Patients. J Clin Med. 2019 Aug 16;8(8):1235. doi: 10.3390/jcm8081235. PMID 31426378
- [Background] Lee JH, Nam S, Jang YE, Kim EH, Kim HS, Kim JT. Clinical performance of Ambu AuraGainTM versus i-gelTM in anesthetized children: a prospective, randomized controlled trial. Anesth Pain Med (Seoul). 2020 Apr 30;15(2):173-180. doi: 10.17085/apm.2020.15.2.173. Epub 2020 Apr 29. PMID 33329810